CLINICAL TRIAL: NCT00671281
Title: The Effect of Tranexamic Acid on Intraoperative and Post-Operative Bleeding in Functional Endoscopic Sinus Surgery: A Randomized, Prospective, Double-Blinded Study
Brief Title: The Effect of Tranexamic Acid on Intraoperative and Post-Operative Bleeding in Functional Endoscopic Sinus Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was cancelled
Sponsor: University of Calgary (Other)
Responsible Party: Dr. Brad Mechor, Division of Otolaryngology, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tranexamic Acid in FESS
Record Dates: First submitted 2008-04-30; First posted 2008-05-05 (Estimated); Last update posted 2010-09-03 (Estimated); Status verified 2010-09

CONDITIONS: Chronic Sinusitis
Keywords: FESS; Tranexamic acid; Hemostasis; Visualization
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- B (Experimental): This group will be the experimental group which will receive tranexamic acid in oral form three days before and six days after surgery.
  Interventions: Drug: Tranexamic acid
- A (Placebo Comparator): This will be the control group which will take the placebo medication for 3 days before and six days after their functional endoscopic sinus surgery (FESS).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic acid — Oral form, 100mg, tid (three times per day), 3 days before/the day of/6 days after the surgery
  Other Names: Cyclokapron
  Arms: B
Drug: Placebo — Placebo, Oral form, three times a day, 3 days before/day of/6 days after surgery
  Arms: A

SUMMARY:
Sinus surgery is a common, day surgery procedure performed by general and subspecialty trained otolaryngologists. In most cases, this is a safe surgery with a low incidence of complications. When there is significant bleeding or enough bleeding to obscure important anatomical landmarks, there is a higher chance of complications. These complications can include blindness, meningitis or cerebrospinal fluid leak. Our hypothesis is that in patients taking oral tranexamic acid three days before surgery and six days after, there will be less intraoperative bleeding, better surgical visualization and less postoperative bleeding events.

ELIGIBILITY:
Inclusion Criteria:

* Chronic sinusitis requiring bilateral functional endoscopic sinus surgery
* Between the ages of 18-65
* Willing to comply with standard followup
* No coagulopathy
* Not pregnant

Exclusion Criteria:

* Pregnant
* On anticoagulants within 3 months of the surgery
* Coagulopathy
* <18 or >65 years of age

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-06 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Intraoperative bleeding amount | During the surgery

SECONDARY OUTCOMES:
Surgical visualization scoring | During the surgery
Postoperative bleeding events | Six days after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Brad D Mechor, MD, Principal Investigator — Division of Otolaryngology, University of Calgary
Locations (1):
- Rockyview General Hospital, Calgary, Alberta, Canada

REFERENCES:
- [Background] Osguthorpe JD. Surgical outcomes in rhinosinusitis: what we know. Otolaryngol Head Neck Surg. 1999 Apr;120(4):451-3. doi: 10.1053/hn.1999.v120.a95228. No abstract available. PMID 10187931
- [Background] Blumenfeld RJ, Skolnik EM. Intracranial complications of sinus disease. Trans Am Acad Ophthalmol Otolaryngol. 1966 Nov-Dec;70(6):899-908. No abstract available. PMID 5971474
- [Background] Clayman GL, Adams GL, Paugh DR, Koopmann CF Jr. Intracranial complications of paranasal sinusitis: a combined institutional review. Laryngoscope. 1991 Mar;101(3):234-9. doi: 10.1288/00005537-199103000-00003. PMID 2000009
- [Background] Morgan PR, Morrison WV. Complications of frontal and ethmoid sinusitis. Laryngoscope. 1980 Apr;90(4):661-6. doi: 10.1288/00005537-198004000-00013. PMID 7359985
- [Background] Cumberworth VL, Sudderick RM, Mackay IS. Major complications of functional endoscopic sinus surgery. Clin Otolaryngol Allied Sci. 1994 Jun;19(3):248-53. doi: 10.1111/j.1365-2273.1994.tb01225.x. PMID 7923850
- [Background] Goldwyn RM. Unexpected bleeding after elective nasal surgery. Ann Plast Surg. 1979 Mar;2(3):201-4. doi: 10.1097/00000637-197903000-00004. PMID 539747
- [Background] Dunn CJ, Goa KL. Tranexamic acid: a review of its use in surgery and other indications. Drugs. 1999 Jun;57(6):1005-32. doi: 10.2165/00003495-199957060-00017. PMID 10400410
- [Background] Yaniv E, Shvero J, Hadar T. Hemostatic effect of tranexamic acid in elective nasal surgery. Am J Rhinol. 2006 Mar-Apr;20(2):227-9. PMID 16686395
- [Background] Fremes SE, Wong BI, Lee E, Mai R, Christakis GT, McLean RF, Goldman BS, Naylor CD. Metaanalysis of prophylactic drug treatment in the prevention of postoperative bleeding. Ann Thorac Surg. 1994 Dec;58(6):1580-8. doi: 10.1016/0003-4975(94)91636-5. PMID 7526811
- [Background] Casati V, Sandrelli L, Speziali G, Calori G, Grasso MA, Spagnolo S. Hemostatic effects of tranexamic acid in elective thoracic aortic surgery: a prospective, randomized, double-blind, placebo-controlled study. J Thorac Cardiovasc Surg. 2002 Jun;123(6):1084-91. doi: 10.1067/mtc.2002.120717. PMID 12063454
- [Background] Wormald PJ, van Renen G, Perks J, Jones JA, Langton-Hewer CD. The effect of the total intravenous anesthesia compared with inhalational anesthesia on the surgical field during endoscopic sinus surgery. Am J Rhinol. 2005 Sep-Oct;19(5):514-20. PMID 16270608